CLINICAL TRIAL: NCT00124319
Title: Epidemiology of Jump-Landing Movements and ACL Injury
Brief Title: Risk Factors for Anterior Cruciate Ligament (ACL) Injury
Status: Completed | Type: Observational
Sponsor: Steve Marshall (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Steve Marshall, Professor of Epidemiology, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: R01AR050461 (NIH); R01AR050461 (NIH); R01AR050461-01A1 (NIH)
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2009-05

CONDITIONS: Knee Injuries; Athletic Injuries
Keywords: Biomechanics; Neuromuscular; Lower limb; Injury; ACL; Anterior Cruciate Ligament injury
MeSH Terms: conditions — Knee Injuries; Athletic Injuries; Wounds and Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Incoming cadets at the U.S. Naval, Air Force, or Military Academies

SUMMARY:
The anterior cruciate ligament (ACL) is located inside the knee joint and provides stability to the knee. ACL injuries occur more frequently in women than men; the reason for this is unknown. The purpose of this study is to determine gender-specific anatomical, hormonal, and demographic risk factors for ACL injury. This observational cohort study will only enroll incoming cadets at the U.S. Naval, Air Force, or Military Academies.

Study hypothesis: Human movement factors, including key kinetics and kinematics of the knee during a jump-landing task, are associated with the rate of ACL injury.

DETAILED DESCRIPTION:
The ACL stabilizes the knee joint by preventing the shinbone (tibia) from sliding forward beneath the thighbone (femur). A hard twist or excessive pressure on the ACL can tear or rupture the ligament, resulting in high levels of short-term disability and extensive rehabilitation. Previous data indicate that women who participate in sports or who are otherwise physically active have higher rates of ACL injury than men; the reason for this is unknown. There are four groups of potential risk factors for ACL injury: environmental, anatomical, hormonal, and biomechanical or neuromuscular. In particular, poor technique when landing from a jump (also known as jump-landing) is proposed as a specific neuromuscular risk factor of interest in this study. This study will determine gender-specific anatomical, hormonal, and demographic risk factors for ACL injury, as well as quantify gender-specific differences in jump-landing technique and other neuromuscular risk factors.

This observational cohort study will enroll 4,800 cadets at the three large U.S. military academies; approximately 50% of those enrolled will be women. Only incoming cadets at the U.S. Naval, Air Force, or Military Academies will be able to participate. Each study participant will undergo a baseline assessment that will include measurement of neuromuscular risk factors using motion analysis, strength testing, and standardized assessment of poor jump-landing technique using the Landing Error Score System (LESS). All participants will be followed for up to 4 years. ACL injuries will be prospectively identified; an injury questionnaire is administered to participants who sustain an ACL injury while they are cadets. Otherwise, there is no further contact.

ELIGIBILITY:
Inclusion Criteria:

* Incoming cadet at the U.S. Naval, Air Force, or Military Academies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Incoming cadets at the U.S. Naval, Air Force, or Military Academies
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2005-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W. Marshall, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - U.S. Air Force Academy, Colorado Springs, Colorado
  - U.S. Naval Academy, Annapolis, Maryland
  - U.S. Military Academy, West Point, New York